CLINICAL TRIAL: NCT02795312
Title: Feasibility, Acceptability and Effectiveness of Modified Mindfulness Based Stress Reduction (MBSR) for Smoking Cessation in Cancer Patients
Brief Title: Mindfulness Based Smoking Cessation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H-34953; 6003740 (Other Grant/Funding Number: Massachusetts Society of Clinical Oncology)
Record Dates: First submitted 2016-06-01; First posted 2016-06-10 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Cancer; Smoking Cessation
Keywords: Cigarette Smoking
MeSH Terms: conditions — Neoplasms; Smoking Cessation; Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smoking Cessation Training Program (Experimental): Participants will take part in a 9-week Smoking Cessation Program class curriculum consisting of weekly 2.5 hour classes and complete pre and post questionnaires
  Interventions: Behavioral: Smoking Cessation Program

INTERVENTIONS:
Behavioral: Smoking Cessation Program — Participants will take part in a 9-week Smoking Cessation Program

SUMMARY:
This is a study designed to mindfulness based stress reduction (MBSR) training program to assess feasibility and acceptability of the intervention. Participants will participate in a 9-week training program and complete pre-and post-questionnaires. Participants will have the option of participating in a follow-up focus group.

DETAILED DESCRIPTION:
The investigators will introduce a mindfulness based stress reduction (MBSR) training program at Boston Medical Center's oncology clinic to promote engagement of low-income and minority smokers with cancer in smoking cessation. This training will follow an adapted MBSR curriculum designed by and for Boston Medical Center patients with chronic pain in the Integrated Medical Group Visit research program in Family Medicine. The investigators will tailor this adapted MBSR curriculum to address smoking cessation. To test the feasibility and acceptability of our intervention, the investigators will pilot test it with 30 patients over the course of three MBSR training programs (each cohort is 9 weeks). The investigators will acquire feasibility data (number of inquiries, number of sessions attended, and satisfaction with MBSR). Additionally, pre and post questionnaires will assess readiness to quit, stress level, and satisfaction with and acceptability of MBSR after every cohort). The primary outcome is engagement in smoking cessation treatment which includes counseling and/or pharmacotherapy. Additionally, the investigators will hold a focus group after each of the 3 cohorts have completed the program to discuss acceptability of study materials as well as facilitators and barriers to participation in the training. Data collected from this study will generate preliminary data to successfully justify and secure future funding for a larger controlled study.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* smoked cigarettes in the past week
* cancer diagnosis more than 6 months
* have a scheduled visit in the oncology clinic with an oncologist or mid-level provider
* telephone access
* English speaking for screening/consenting purposes
* able and willing to participate in the study protocol and provide informed consent

Exclusion Criteria:

* cancer prognosis less than 6 months
* planning to move out of the area within 6 months
* actively using evidence-based smoking cessation treatment during screening
* pregnant women and women planning on becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Number of participants engaged in smoking cessation counseling | 3 months
  Participants will complete a weekly intake form and a telephone based questionnaire at 3 months to assess engagement in evidence based smoking cessation counseling by completion of one of the following: (a) at least 1 visit with Boston Medical Center pulmonary smoking cessation program for individual quit plan, or (b) at least 1 telephone based Quitworks counseling session, or (c) >1 PCP or Oncology visit in which smoking cessation treatment is discussed.

SECONDARY OUTCOMES:
Number of patients with reduced stress assessed using validated Perceived Stress Scale (PSS) | 3 months
  Stress reduction will be assessed using validated Perceived Stress Scale (PSS)
Number of patients reporting readiness to quit smoking based on the Transtheoretical Model and Stages of Change | 3 months
  Patient self report of readiness to quit smoking based on stage of change: precontemplation, contemplation, preparation or action assessed on questionnaire at baseline, 9 weeks, and at 3 month follow up
Number of participants identifying a smoking quit date | 3 months
  Participant will report if quit date has been determined on weekly questionnaire and/or at three month follow up
Number of participants reporting 7 day smoking abstinence from cigarettes | 3 months
  Participant will report 7 day smoking abstinence from cigarettes on weekly questionnaire and/or at three month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Marjory Charlot, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be included in any publications